CLINICAL TRIAL: NCT02579265
Title: A Prospective, Randomized, Controlled, Double-Blind, Parallel-Group, Phase 3 Study to Compare Safety and Efficacy of Smoflipid 20% to Intralipid 20% in Hospitalized Neonates and Infants Requiring 28 Days of Parenteral Nutrition
Brief Title: Phase 3 Study to Compare Safety and Efficacy of Smoflipid 20% to Intralipid 20% in Hospitalized Neonates and Infants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Outcome of a planned interim analysis was that the sample size required to show superiority was too high to be feasible. Fresenius Kabi requested termination to the FDA on 17 Jan 2020. FDA accepted termination by written response on 16 Apr 2020.
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SMOF-018-CP3
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Hospitalized Neonates and Infants, Expected to Require Parenteral Nutrition for 28 Days
Keywords: Parenteral nutrition; Neonates; Infants; Lipid emulsions; Intravenous
MeSH Terms: conditions — Hyperphagia | interventions — SMOFlipid; Parenteral Nutrition; soybean oil, phospholipid emulsion; Fat Emulsions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoflipid 20% (Experimental): Smoflipid is a lipid emulsion containing soybean oil, MCTs (medium-chain triglycerides), olive oil, and fish oil. Smoflipid belongs to the pharmacotherapeutic group: "Solutions for parenteral nutrition, fat emulsions".
  Interventions: Drug: Smoflipid 20% (investigational lipid for parenteral nutrition)
- Intralipid® 20% (Active Comparator): Intralipid is a long-chain triglyceride emulsion derived from purified soybean oil and egg yolk phospholipids. Intralipid belongs to the pharmacotherapeutic group: "Solutions for parenteral nutrition, fat emulsions".
  Interventions: Drug: Intralipid® 20%

INTERVENTIONS:
Drug: Smoflipid 20% (investigational lipid for parenteral nutrition) — Dose: The targeted maximal dose is 3.0 g/kg/day. In patients already receiving parenteral nutrition (PN) before starting study treatment, the dose will either stay at 3.0 g/kg/day or be increased by 1.0 g/kg/day steps to a maximum of 3.0 g/kg/day.
  Smoflipid 20% will be infused over 20 - 24 hours, as per hospital policy, at a weight based infusion rate.
  Smoflipid 20% will be infused into a central or a peripheral vein.
  Other Names: Smoflipid 20% (lipid injectable emulsion)
  Arms: Smoflipid 20%
Drug: Intralipid® 20% — Dose: The targeted maximal dose is 3.0 g/kg/day. In patients already receiving parenteral nutrition (PN) before starting study treatment, the dose will either stay at 3.0 g/kg/day or be increased by 1.0 g/kg/day steps to a maximum of 3.0 g/kg/day.
  Intralipid® 20% will be infused over 20 - 24 hours, as per hospital policy, at a weight based infusion rate.
  Intralipid® 20% will be infused into a central or peripheral vein.
  Other Names: Intralipid® 20% (a 20% intravenous fat emulsion)
  Arms: Intralipid® 20%

SUMMARY:
To show the superiority in safety of Smoflipid over Intralipid® as measured by the number of study patients in each treatment group with conjugated bilirubin exceeding 2 mg/dL during the first 28 days of study treatment, confirmed by a second sample collected 7 days after the first sample.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants, expected to require parenteral nutrition (PN) for 28 days
* Postmenstrual age ≥ 24 weeks
* Birth weight ≥ 750g
* Gastroschisis, duodenal, jejunal or ileal atresia, volvulus, spontaneous intestinal perforation or necrotizing enterocolitis (Bell's stage 2B or higher)
* At least 80% of nutritional needs at baseline received by PN
* Signed and dated informed consent obtained from at least one parent or legal guardian

Exclusion Criteria:

* Conjugated bilirubin > 0.6 mg/dL
* Any known pre-, intra- or posthepatic complication increasing conjugated bilirubin levels > 0.6, mg/dL during study participation
* Suspected liver disease or liver damage based on either aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyl transferase (GGT) exceeding 2.5x upper limit of normal range
* Active bloodstream infection demonstrated by positive blood culture at screening
* Cystic fibrosis
* Meconium ileus
* Serum triglyceride levels > 250 mg/dL
* Cyanotic congenital heart defect
* Severe renal failure with serum creatinine > 2.0 mg/dL
* History of shock requiring vasopressors
* Anasarca
* Extracorporeal Membrane Oxygenation (ECMO)
* Known inborn errors of metabolism
* Known congenital viral infection
* Unlikely to survive longer than 28 days
* Known hypersensitivity to fish-, egg-, soya- or peanut protein or to any of the active substances or excipients

Min Age: 0 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Abrams, MD, Principal Investigator — University of Texas at Austin
Locations (13):
- United States (13):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - UC San Diego Medical Center, San Diego, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Yale - New Haven Children's Hospital, New Haven, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Steven & Alexandra Cohen Children's Medical Center of NY, New York, New York
  - The Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Abrams SA, Ernst KD, Weitkamp JH, Mascarenhas M, Anderson-Berry A, Rudolph J, Ling CY, Robinson DT, Shores D, Hair AB, Lai J, Lane B, McCallie KR, Levit O, Kim JH. Safety and Efficacy of a Composite Lipid Emulsion with Fish Oil in Hospitalized Neonates and Infants Requiring Prolonged Parenteral Nutrition - A Randomized, Double-Blind, Multicenter, Controlled Trial. J Nutr. 2024 Dec;154(12):3615-3625. doi: 10.1016/j.tjnut.2024.10.005. Epub 2024 Oct 5. PMID 39374788

RESULTS

PARTICIPANT FLOW:
Groups:
- Smoflipid 20%: Smoflipid is a lipid emulsion containing soybean oil, MCTs (medium-chain triglycerides), olive oil, and fish oil. Smoflipid belongs to the pharmacotherapeutic group: "Solutions for parenteral nutrition, fat emulsions".
  Smoflipid 20% (investigational lipid for parenteral nutrition): Dose: The targeted maximal dose is 3.0 g/kg/day.
  In patients already receiving parenteral nutrition (PN) before starting study treatment, the dose will either stay at 3.0 g/kg/day or be increased by 1.0 g/kg/day steps to a maximum of 3.0 g/kg/day.
  Smoflipid 20% will be infused over 20 - 24 hours, as per hospital policy, at a weight based infusion rate.
  Smoflipid 20% will be infused into a central or a peripheral vein.
- Intralipid® 20%: Intralipid is a long-chain triglyceride emulsion derived from purified soybean oil and egg yolk phospholipids. Intralipid belongs to the pharmacotherapeutic group: "Solutions for parenteral nutrition, fat emulsions".
  Intralipid® 20%: Dose: The targeted maximal dose is 3.0 g/kg/day. In patients already receiving parenteral nutrition (PN) before starting study treatment, the dose will either stay at 3.0 g/kg/day or be increased by 1.0 g/kg/day steps to a maximum of 3.0 g/kg/day.
  Intralipid® 20% will be infused over 20 - 24 hours, as per hospital policy, at a weight based infusion rate.
  Intralipid® 20% will be infused into a central or peripheral vein.
Period: Overall Study
Arm/Group | Smoflipid 20% | Intralipid® 20%
Started | 83 | 78
Completed | 33 | 33
Not Completed | 50 | 45
Not completed — Weaned off earlier than 28 days | 44 | 43
Not completed — Adverse Event | 2 | 0
Not completed — Any other reason not specified | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal due to increased conjugated bilirubin | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intralipid® 20% | Smoflipid 20% | Total
Number analyzed (Participants) | 78 | 83 | 161
Age, Continuous [Mean (Standard Deviation); unit: days] | 8.3 (12.16) | 11.4 (21.58) | 9.9 (17.67)
Age, Customized [Count of Participants; unit: Participants]
  Age category: Newborn (0-27 days) | 75 | 77 | 152
  Age category: Infant (>=28 days) | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 84
  Male | 33 | 44 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 17 | 25
  Not Hispanic or Latino | 70 | 66 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 4 | 15
  White | 57 | 65 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 10 | 16
Postmenstrual age at birth [Mean (Standard Deviation); unit: days] | 238.4 (23.98) | 243.2 (24.27) | 240.9 (24.18)
Underlying disease type [Count of Participants; unit: Participants]
  No NEC | 72 | 74 | 146
  NEC | 6 | 9 | 15
Body weight [Mean (Standard Deviation); unit: kg] — Population: Missing
  kg
    number analyzed (Participants) | 74 | 82 | 156
    (all) | 2.25 (0.663) | 2.44 (0.871) | 2.35 (0.783)
Body weight Z-score [Mean (Standard Deviation); unit: units on a scale] — Z-scores are used to display and interpret growth measurements. In childhood, sex and age-adjusted Z-scores for weight, height, and head circumference are routinely used to assess growth and nutritional status - They are derived by comparing individual growth measurements against growth charts from a 'normal' population. Z-score is the distance and direction of an observation away from the 'normal' population mean (Z-score=0).
  Z-scores <=2 indicate:
  Underweight (for body weight assessment) Stunted (for body length assessment) Microcephaly (for head circumference assessment)
  units on a scale | -0.90 (0.969) | -1.06 (1.090) | -0.98 (1.034)
Body weight (category for age) [Count of Participants; unit: Participants] — Population: Missing
  Data were age-standardized using growth charts as suggested by Fenton (Fenton et al., 2013) and the World Health Organization (WHO) Multicenter Growth Reference Study (MGRS; WHO 2006, 2007).
  Participants
    number analyzed (Participants) | 74 | 82 | 156
    Low | 12 | 20 | 32
    Normal | 62 | 62 | 124
    High | 0 | 0 | 0
Body length [Mean (Standard Deviation); unit: cm] — Population: Missing
  cm
    number analyzed (Participants) | 72 | 78 | 150
    (all) | 44.36 (4.407) | 45.15 (5.024) | 44.77 (4.739)
Body length Z-score [Mean (Standard Deviation); unit: units on a scale] — Z-scores are used to display and interpret growth measurements. In childhood, sex and age-adjusted Z-scores for weight, height, and head circumference are routinely used to assess growth and nutritional status - They are derived by comparing individual growth measurements against growth charts from a 'normal' population. Z-score is the distance and direction of an observation away from the 'normal' population mean (Z-score=0).
  Z-scores <=2 indicate:
  Underweight (for body weight assessment) Stunted (for body length assessment) Microcephaly (for head circumference assessment) Population: Missing
  units on a scale
    number analyzed (Participants) | 72 | 78 | 150
    (all) | -1.02 (1.124) | -1.21 (1.339) | -1.11 (1.240)
Body length (category for age) [Count of Participants; unit: Participants] — Population: Missing
  Data were age-standardized using growth charts as suggested by Fenton (Fenton et al., 2013) and the World Health Organization (WHO) Multicenter Growth Reference Study (MGRS; WHO 2006, 2007).
  Participants
    number analyzed (Participants) | 72 | 78 | 150
    Low | 12 | 25 | 37
    Normal | 60 | 53 | 113
    High | 0 | 0 | 0
Head circumference [Mean (Standard Deviation); unit: cm] — Population: Missing
  cm
    number analyzed (Participants) | 73 | 78 | 151
    (all) | 31.28 (2.798) | 31.69 (3.225) | 31.49 (3.024)
Head circumference Z-score [Mean (Standard Deviation); unit: units on a scale] — Z-scores are used to display and interpret growth measurements. In childhood, sex and age-adjusted Z-scores for weight, height, and head circumference are routinely used to assess growth and nutritional status - They are derived by comparing individual growth measurements against growth charts from a 'normal' population. Z-score is the distance and direction of an observation away from the 'normal' population mean (Z-score=0).
  Z-scores <=2 indicate:
  Underweight (for body weight assessment) Stunted (for body length assessment) Microcephaly (for head circumference assessment) Population: Missing
  units on a scale
    number analyzed (Participants) | 73 | 78 | 151
    (all) | -0.76 (1.184) | -0.97 (1.249) | -0.87 (1.218)
Head circumference (category for age) [Count of Participants; unit: Participants] — Population: Missing
  Data were age-standardized using growth charts as suggested by Fenton (Fenton et al., 2013) and the World Health Organization (WHO) Multicenter Growth Reference Study (MGRS; WHO 2006, 2007).
  Participants
    number analyzed (Participants) | 73 | 78 | 151
    Low | 9 | 20 | 29
    Normal | 62 | 57 | 119
    High | 2 | 1 | 3
Duration of pretreatment [Mean (Standard Deviation); unit: days] — Population: Missing
  days
    number analyzed (Participants) | 45 | 49 | 94
    (all) | 8.8 (8.25) | 7.3 (7.50) | 8.0 (7.86)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in Each Treatment Group With Conjugated Bilirubin Levels > 2 mg/dL During the First 28 Days of Study Treatment, Confirmed by a Second Sample Collected 7 Days After the First Sample
Description: Analysis of patients with Event at any timepoint of sampling (i.e. Day 8, 15, 22, 29/end of Treatment) and subsequent (i.e. +7 days) confirmation.
Time Frame: Screening, Day 8, 15, 22, 29/end of treatment + confirmatory sample: 7 days after conjugated bilirubin level exceeds 2 mg/dl
Population: The numbers in the subgroups refer to 100%
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Combined | 3 | 2
  NEC: number analyzed (Participants) | 6 | 9
  NEC | 0 | 1
  No NEC: number analyzed (Participants) | 72 | 74
  No NEC | 3 | 1

2. Secondary Outcome: Body Weight (Change From Baseline)
Description: Data were age-standardized using growth charts as suggested by Fenton (Fenton et al., 2013) and the World Health Organization (WHO) Multicenter Growth Reference Study (MGRS; WHO 2006, 2007).
Time Frame: Day 1-29, and at Follow-up (+7 days) (if continued: until Day 85 + at Follow up)
Population: The numbers at different timepoints refer to 100%. Timepoints >10% of Subjects (overall) are displayed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Baseline: number analyzed (Participants) | 74 | 82
  Baseline: Low | 12 | 20
  Baseline: Normal | 62 | 62
  Baseline: High | 0 | 0
  Day 8: number analyzed (Participants) | 76 | 77
  Day 8: Low | 14 | 22
  Day 8: Normal | 61 | 55
  Day 8: High | 1 | 0
  Day 15: number analyzed (Participants) | 58 | 64
  Day 15: Low | 13 | 16
  Day 15: Normal | 45 | 48
  Day 15: High | 0 | 0
  Day 22: number analyzed (Participants) | 39 | 45
  Day 22: Low | 8 | 14
  Day 22: Normal | 31 | 31
  Day 22: High | 0 | 0
  Day 29: number analyzed (Participants) | 31 | 33
  Day 29: Low | 6 | 9
  Day 29: Normal | 25 | 24
  Day 29: High | 0 | 0
  Day 36: number analyzed (Participants) | 21 | 18
  Day 36: Low | 4 | 5
  Day 36: Normal | 16 | 13
  Day 36: High | 1 | 0
  Day 43: number analyzed (Participants) | 17 | 12
  Day 43: Low | 2 | 3
  Day 43: Normal | 15 | 8
  Day 43: High | 0 | 1
  Day 50: number analyzed (Participants) | 12 | 10
  Day 50: Low | 2 | 3
  Day 50: Normal | 10 | 7
  Day 50: High | 0 | 0
  Day 57: number analyzed (Participants) | 11 | 8
  Day 57: Low | 1 | 1
  Day 57: Normal | 10 | 7
  Day 57: High | 0 | 0
  Day 64: number analyzed (Participants) | 9 | 6
  Day 64: Low | 0 | 0
  Day 64: Normal | 9 | 6
  Day 64: High | 0 | 0
  Follow-up: number analyzed (Participants) | 60 | 55
  Follow-up: Low | 16 | 15
  Follow-up: Normal | 43 | 40
  Follow-up: High | 1 | 0

3. Secondary Outcome: Body Length (Change From Baseline)
Description: as for outcome 2
Time Frame: Day 1, 8, 15, 22, 29/end of treatment, if continued: Day 36, 43, 50, 57, 64, 71, 78, 85/end of treatment, Follow-up
Population: The numbers at different timepoints refer to 100%. Timepoints >10% of Subjects (overall) are displayed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Baseline: number analyzed (Participants) | 72 | 78
  Baseline: Low | 12 | 25
  Baseline: Normal | 60 | 53
  Baseline: High | 0 | 0
  Day 8: number analyzed (Participants) | 73 | 79
  Day 8: Low | 14 | 30
  Day 8: Normal | 59 | 49
  Day 8: High | 0 | 0
  Day 15: number analyzed (Participants) | 61 | 64
  Day 15: Low | 14 | 25
  Day 15: Normal | 47 | 39
  Day 15: High | 0 | 0
  Day 22: number analyzed (Participants) | 41 | 46
  Day 22: Low | 10 | 17
  Day 22: Normal | 31 | 29
  Day 22: High | 0 | 0
  Day 29: number analyzed (Participants) | 33 | 33
  Day 29: Low | 6 | 13
  Day 29: Normal | 27 | 20
  Day 29: High | 0 | 0
  Day 36: number analyzed (Participants) | 21 | 16
  Day 36: Low | 7 | 6
  Day 36: Normal | 14 | 10
  Day 36: High | 0 | 0
  Day 43: number analyzed (Participants) | 17 | 13
  Day 43: Low | 4 | 4
  Day 43: Normal | 13 | 9
  Day 43: High | 0 | 0
  Day 50: number analyzed (Participants) | 15 | 10
  Day 50: Low | 5 | 2
  Day 50: Normal | 10 | 8
  Day 50: High | 0 | 0
  Day 57: number analyzed (Participants) | 11 | 8
  Day 57: Low | 1 | 1
  Day 57: Normal | 9 | 6
  Day 57: High | 1 | 1
  Follow up: number analyzed (Participants) | 56 | 53
  Follow up: Low | 16 | 26
  Follow up: Normal | 40 | 27
  Follow up: High | 0 | 0

4. Secondary Outcome: Head Circumference (Change From Baseline)
Description: as for outcome 2
Time Frame: Day 1, 8, 15, 22, 29/end of treatment, if continued: Day 36, 43, 50, 57, 64, 71, 78, 85/end of treatment, Follow-up
Population: The numbers at different timepoints refer to 100%. Timepoints >10% of Subjects (overall) are displayed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Baseline: number analyzed (Participants) | 73 | 78
  Baseline: Low | 9 | 20
  Baseline: Normal | 62 | 57
  Baseline: High | 2 | 1
  Day 8: number analyzed (Participants) | 73 | 81
  Day 8: Low | 10 | 21
  Day 8: Normal | 63 | 59
  Day 8: High | 0 | 1
  Day 15: number analyzed (Participants) | 61 | 65
  Day 15: Low | 7 | 13
  Day 15: Normal | 54 | 51
  Day 15: High | 0 | 1
  Day 22: number analyzed (Participants) | 41 | 46
  Day 22: Low | 5 | 12
  Day 22: Normal | 36 | 34
  Day 22: High | 0 | 0
  Day 29: number analyzed (Participants) | 33 | 33
  Day 29: Low | 3 | 8
  Day 29: Normal | 30 | 25
  Day 29: High | 0 | 0
  Day 36: number analyzed (Participants) | 20 | 16
  Day 36: Low | 2 | 5
  Day 36: Normal | 18 | 10
  Day 36: High | 0 | 1
  Day 43: number analyzed (Participants) | 17 | 13
  Day 43: Low | 1 | 2
  Day 43: Normal | 16 | 11
  Day 43: High | 0 | 0
  Day 50: number analyzed (Participants) | 15 | 10
  Day 50: Low | 1 | 1
  Day 50: Normal | 14 | 8
  Day 50: High | 0 | 1
  Day 57: number analyzed (Participants) | 9 | 7
  Day 57: Low | 0 | 0
  Day 57: Normal | 9 | 6
  Day 57: High | 0 | 1
  Day 64: number analyzed (Participants) | 8 | 5
  Day 64: Low | 0 | 0
  Day 64: Normal | 8 | 5
  Day 64: High | 0 | 0
  Follow up: number analyzed (Participants) | 55 | 51
  Follow up: Low | 9 | 9
  Follow up: Normal | 46 | 39
  Follow up: High | 0 | 3

5. Secondary Outcome: Time to Full Enteral or Oral Feeds
Description: Time to full enteral or oral feeds (i.e. PN weaning) is the time from the randomization date to the date of the first full enteral or oral Feeds.
Time Frame: Day 29/end of treatment, if continued: Day 85/end of treatment
Population: The Standard Deviation for Time to Event was not calculated. NA=Not available
Measure: Median (95% Confidence Interval); unit: Time to event in days
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 58 | 58
Time to event in days | 21.95 [NA to NA] — The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach. | 23.29 [NA to NA] — The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach.

6. Secondary Outcome: Fatty Acids in Plasma and Red Blood Cell Membranes (Change From Baseline)
Description: RBC refers to red blood cells. Timepoints >10% of Subjects (overall) are displayed.
Time Frame: Day 1, Day 29/end of treatment, if continued: Day 57, 85/end of treatment
Population: Over time analysis of laboratory parameters were assessed at all timepoints as available
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 70 | 78
ug/mL
  Eicosapentaenoic acid Baseline | 7.36 (6.545) | 14.52 (16.480)
  Eicosapentaenoic acid Change to EoT: number analyzed (Participants) | 60 | 69
  Eicosapentaenoic acid Change to EoT | -1.57 (7.336) | 30.44 (38.615)
  Eicosapentaenoic acid Change to EoT extension phase: number analyzed (Participants) | 11 | 12
  Eicosapentaenoic acid Change to EoT extension phase | 1.96 (10.389) | 40.62 (51.417)
  Docosahexaenoic acid Baseline | 41.14 (14.724) | 47.31 (18.484)
  Docosahexaenoic Acid Change to Eot: number analyzed (Participants) | 60 | 69
  Docosahexaenoic Acid Change to Eot | -1.36 (17.721) | 40.06 (28.678)
  Docosahexaenoic Acid Change to EoT extension: number analyzed (Participants) | 11 | 12
  Docosahexaenoic Acid Change to EoT extension | 9.55 (19.462) | 49.93 (41.868)
  Arachidonic Acid Baseline | 148.80 (52.531) | 149.42 (47.438)
  Arachidonic Acid Change to EoT: number analyzed (Participants) | 60 | 69
  Arachidonic Acid Change to EoT | -25.36 (59.925) | -31.47 (54.249)
  Arachidonic Acid Change to EoT extension: number analyzed (Participants) | 11 | 12
  Arachidonic Acid Change to EoT extension | -8.18 (51.138) | -60.00 (73.737)
  Alpha-linolenic Acid Baseline: number analyzed (Participants) | 68 | 78
  Alpha-linolenic Acid Baseline | 19.24 (12.675) | 16.57 (13.081)
  Alpha-linolenic Acid Change to EoT: number analyzed (Participants) | 58 | 69
  Alpha-linolenic Acid Change to EoT | -2.01 (17.452) | -3.31 (13.250)
  Alpha-linolenic Acid Change to EoT extension: number analyzed (Participants) | 9 | 12
  Alpha-linolenic Acid Change to EoT extension | 5.88 (19.477) | -0.55 (11.454)
  Linoleic acid Baseline | 460.62 (211.354) | 427.44 (185.206)
  Linoleic acid Change to EoT: number analyzed (Participants) | 60 | 69
  Linoleic acid Change to EoT | 50.95 (270.029) | -41.68 (190.749)
  Linoleic acid Change to EoT extension: number analyzed (Participants) | 11 | 12
  Linoleic acid Change to EoT extension | 209.99 (286.361) | -50.25 (2011.292)
  Mead acid Baseline | 4.42 (5.888) | 4.35 (7.620)
  Mead acid Change to EoT: number analyzed (Participants) | 60 | 69
  Mead acid Change to EoT | -2.46 (6.816) | -2.19 (8.011)
  Mead Acid Change to EoT extension: number analyzed (Participants) | 11 | 12
  Mead Acid Change to EoT extension | 1.82 (9.045) | -6.94 (17.595)
  RBC Eicosapentaenoic acid Baseline: number analyzed (Participants) | 68 | 74
  RBC Eicosapentaenoic acid Baseline | 4.20 (2.533) | 5.21 (3.954)
  RBC Eicosapentaenoic acid Change to EoT: number analyzed (Participants) | 54 | 64
  RBC Eicosapentaenoic acid Change to EoT | 0.56 (2.375) | 19.22 (11.433)
  RBC Eicosapentaenoic acid Change to EoT extension: number analyzed (Participants) | 10 | 12
  RBC Eicosapentaenoic acid Change to EoT extension | 2.05 (2.841) | 31.83 (11.973)
  RBC Docosahexaenoic acid Baseline: number analyzed (Participants) | 69 | 76
  RBC Docosahexaenoic acid Baseline | 94.18 (26.246) | 92.53 (28.435)
  RBC Docosahexaenoic acid Change to EoT: number analyzed (Participants) | 55 | 65
  RBC Docosahexaenoic acid Change to EoT | -41.60 (53.983) | -40.92 (60.930)
  RBC Docosahexaenoic acid Change to EoT extension: number analyzed (Participants) | 10 | 12
  RBC Docosahexaenoic acid Change to EoT extension | -15.81 (22.577) | 34.85 (17.145)
  RBC Arachidonic acid Baseline: number analyzed (Participants) | 69 | 76
  RBC Arachidonic acid Baseline | 281.53 (63.839) | 268.99 (71.369)
  RBC Arachidonic acid Change to EoT: number analyzed (Participants) | 55 | 65
  RBC Arachidonic acid Change to EoT | -41.60 (53.983) | -40.92 (60.930)
  RBC Arachidonic acid Change to EoT extension: number analyzed (Participants) | 10 | 12
  RBC Arachidonic acid Change to EoT extension | -47.30 (62.470) | -66.75 (47.096)
  RBC Alpha-linolenic acid Baseline: number analyzed (Participants) | 65 | 72
  RBC Alpha-linolenic acid Baseline | 2.31 (1.014) | 2.12 (1.060)
  RBC Alpha-linolenic acid Change to EoT: number analyzed (Participants) | 51 | 61
  RBC Alpha-linolenic acid Change to EoT | 0.52 (1.312) | -0.04 (1.049)
  RBC Alpha-linolenic acid Change to EoT extension: number analyzed (Participants) | 8 | 11
  RBC Alpha-linolenic acid Change to EoT extension | 1.37 (0.587) | -0.17 (1.365)
  RBC Linoleic acid Baseline: number analyzed (Participants) | 69 | 76
  RBC Linoleic acid Baseline | 140.45 (57.461) | 130.67 (53.022)
  RBC Linoleic acid Change to EoT: number analyzed (Participants) | 55 | 65
  RBC Linoleic acid Change to EoT | 57.04 (64.201) | 4.29 (42.276)
  RBC Linoleic acid Change to EoT extension: number analyzed (Participants) | 10 | 12
  RBC Linoleic acid Change to EoT extension | 86.36 (77.716) | 0.06 (68.506)
  RBC Mead acid Baseline: number analyzed (Participants) | 63 | 73
  RBC Mead acid Baseline | 9.21 (4.378) | 8.30 (4.289)
  RBC Mead acid Change to EoT: number analyzed (Participants) | 49 | 63
  RBC Mead acid Change to EoT | -4.19 (3.315) | -3.50 (2.872)
  RBC Mead acid Change to EoT extension: number analyzed (Participants) | 10 | 10
  RBC Mead acid Change to EoT extension | -7.45 (4.576) | -5.40 (3.777)

7. Secondary Outcome: Length of Stay in Hospital
Description: Length of stay in hospital (time from randomization to discharge) was be calculated.
  NA=Not available
Time Frame: Day 1- Follow up (7 days after end of treatment)
Measure: Median (95% Confidence Interval); unit: Median time (days) until discharge
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 61 | 58
Median time (days) until discharge | 65.0 [NA to NA] — The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach. | 50.5 [NA to NA] — The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach.

8. Secondary Outcome: Ratio of Independent Bloodstream Infections to Number of Days on Study Medication
Description: The Ratio is the incidence of bloodstream infection by numbers of day on study medication.
Time Frame: Day 1-29 or -85 if continued + Follow-up
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
ratio | 0.002 (0.0105) | 0.003 (0.0123)

9. Secondary Outcome: Number of Patients With 1 or More Bloodstream Infections to Number of Patients on Study Medication
Time Frame: Day 1-29 or -85 if continued + Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants | 5 | 6

10. Secondary Outcome: Number of Patients Who Complete PN Treatment Without Lipid Minimization
Description: The Analysis was conducted over all study phases.
Time Frame: Day 1-29 or -85 if continued + Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants | 73 | 79

11. Secondary Outcome: Number of Patients Needing to be Withdrawn From the Study Due to Elevated Conjugated Bilirubin Levels
Time Frame: Day 1-29 or -85 if continued + Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Initial Treatment Phase | 0 | 1
  Extension Phase | 0 | 0

12. Secondary Outcome: Area Under the Curve for Time Period in Which Conjugated Bilirubin Levels Are > 1.5 mg/dL in Patients Who Are Not Withdrawn From the Study
Description: The area under the curve (AUC>1.5) is defined as the area between conjugated bilirubin concentrations > 1.5 mg/dL and the horizontal line at 1.5 mg/dL, restricted by the time point of study withdrawal, if applicable. Analysis displays the summary of Area Under the Curve of Bilirubin Levels for the Time Period in Which Conjugated are >1.5 mg/dL
Time Frame: Day 1-29 or -85 if continued + Follow-up
Population: Missing
Measure: Mean (Standard Deviation); unit: mg/dl*days
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
mg/dl*days
  Initial Treatment Phase: number analyzed (Participants) | 66 | 68
  Initial Treatment Phase | 0.587 (2.6620) | 0.804 (3.4700)
  Extended Treatment Phase: number analyzed (Participants) | 11 | 5
  Extended Treatment Phase | 11.609 (15.184) | 0.900 (2.013)

13. Secondary Outcome: Cumulative Number of Days Patients Are Administered a Lipid Dose Without Lipid Minimization
Description: The Analysis was performed over the entire study period.
Time Frame: Day 1-29 or -85 if continued + Follow-up
Population: Missing
Measure: Mean (Standard Deviation); unit: Cumulative days
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 73 | 79
Cumulative days | 27.8 (21.98) | 26.7 (19.94)

14. Secondary Outcome: Time to Conjugated Bilirubin > 2 mg/dL (Confirmed by a Second Sample Collected 7 Days After the First)
Time Frame: Day 1-29 or -85 if continued + Follow-up
Population: NA=Not available Since the number of events was not sufficient, no further analysis was performed.
Measure: Mean (95% Confidence Interval); unit: Number of days
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Number of days | NA [NA to NA] — Not calculated due to due to low number of Events. The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach. | NA [NA to NA] — Not calculated due to due to low number of Events. The cumulative incidence function for competing events (refer to Austin et al. Circulation. 2016 Feb 9; 133(6): 601-609) was used for the interpolation of the median time to event. 95% CIs were not calculated due to this approach.

15. Secondary Outcome: Blood Sampling for Special Analysis (Sterols Including Phytosterols, α-tocopherol)
Time Frame: Day 1, Day 29/end of treatment, if continued: Day 57, 85/end of treatment
Population: Over time analysis of laboratory parameters were assessed at all timepoints as available. Timepoints >10% of Subjects (overall) are displayed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 70 | 78
ug/mL
  Beta(b-) sitosterol Baseline | 45.076 (28.8520) | 41.900 (28.7879)
  b-sitosterol Change to EoT: number analyzed (Participants) | 59 | 69
  b-sitosterol Change to EoT | 39.854 (38.5996) | -6.357 (22.4175)
  b-sitosterol Change to EoT extension: number analyzed (Participants) | 10 | 12
  b-sitosterol Change to EoT extension | 129.938 (52.8942) | -14.247 (46.0845)
  Campesterol Baseline: number analyzed (Participants) | 70 | 77
  Campesterol Baseline | 12.396 (10.1990) | 11.628 (10.4005)
  Campesterol Change to EoT: number analyzed (Participants) | 60 | 69
  Campesterol Change to EoT | 15.385 (21.4772) | -3.079 (9.6125)
  Campesterol Change to EoT extension: number analyzed (Participants) | 10 | 12
  Campesterol Change to EoT extension | 56.681 (34.4784) | -8.159 (22.0449)
  Stigmasterol Baseline: number analyzed (Participants) | 66 | 72
  Stigmasterol Baseline | 7.649 (4.0597) | 6.473 (3.5595)
  Stigmasterol Change to EoT: number analyzed (Participants) | 54 | 63
  Stigmasterol Change to EoT | 4.830 (5.6464) | -2.658 (3.2875)
  Stigmasterol Change to EoT extension: number analyzed (Participants) | 8 | 11
  Stigmasterol Change to EoT extension | 17.862 (3.0202) | -2.422 (5.1974)
  Sitostanol Baseline | 0.838 (0.5692) | 0.710 (0.4423)
  Sitostanol Change to EoT: number analyzed (Participants) | 60 | 69
  Sitostanol Change to EoT | 0.945 (0.9989) | -0.238 (0.4344)
  Sitostanol Change to Eot extension: number analyzed (Participants) | 6 | 6
  Sitostanol Change to Eot extension | 0.134 (0.0931) | -0.169 (0.2486)
  Ergosterol Baseline: number analyzed (Participants) | 40 | 40
  Ergosterol Baseline | 0.028 (0.0210) | 0.025 (0.0215)
  Ergosterol Change to EoT: number analyzed (Participants) | 35 | 38
  Ergosterol Change to EoT | -0.007 (0.0183) | 0.001 (0.0214)
  Ergosterol Change to EoT extension: number analyzed (Participants) | 8 | 8
  Ergosterol Change to EoT extension | 0.002 (0.0038) | -0.010 (0.0267)
  Lathosterol Baseline: number analyzed (Participants) | 65 | 75
  Lathosterol Baseline | 2.411 (0.9417) | 2.215 (1.0751)
  Lathosterol Change to EoT: number analyzed (Participants) | 56 | 62
  Lathosterol Change to EoT | -0.366 (1.1811) | -0.279 (1.1651)
  Lathosterol Change to EoT extension: number analyzed (Participants) | 10 | 12
  Lathosterol Change to EoT extension | -0.801 (0.8797) | -0.956 (2.2253)
  Lanosterol Baseline: number analyzed (Participants) | 65 | 73
  Lanosterol Baseline | 1.281 (0.8046) | 1.135 (0.5630)
  Lanosterol Change to EoT: number analyzed (Participants) | 56 | 60
  Lanosterol Change to EoT | 0.273 (1.0466) | -0.385 (0.5471)
  Lanosterol Change to EoT extension: number analyzed (Participants) | 10 | 12
  Lanosterol Change to EoT extension | 1.039 (0.9342) | -0.548 (0.7836)
  Desmosterol Baseline: number analyzed (Participants) | 64 | 70
  Desmosterol Baseline | 1.396 (1.18371) | 1.196 (1.0923)
  Desmosterol Change to EoT: number analyzed (Participants) | 53 | 59
  Desmosterol Change to EoT | -0.508 (2.0678) | -0.014 (1.3948)
  Desmosterol Change to EoT extension: number analyzed (Participants) | 9 | 11
  Desmosterol Change to EoT extension | -2.337 (4.2890) | -0.562 (1.6695)
  Cholesterol Baseline: number analyzed (Participants) | 69 | 78
  Cholesterol Baseline | 1159.638 (293.2282) | 1163.654 (334.7942)
  Cholesterol Change to EoT: number analyzed (Participants) | 60 | 69
  Cholesterol Change to EoT | -129.433 (295.6223) | -23.072 (358.8932)
  Cholesterol Change to EoT extension: number analyzed (Participants) | 10 | 12
  Cholesterol Change to EoT extension | 145.100 (243.1133) | -232.250 (621.2414)

16. Secondary Outcome: Holman Index
Description: Essential fatty acid deficiency is based on the ratio of Mead acid and Arachidonic acid (also called the triene/tetraene ratio or Holman index; Holman, 1960). A ratio of > 0.2 was considered abnormal (=essential fatty acid deficiency; Holman et al., 1979). Timepoints with >10% of patients are displayed.
Time Frame: Day 1, Day 29/end of treatment, if continued: Day 57, 85/end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid® 20% | Smoflipid 20%
Number analyzed (Participants) | 78 | 83
Participants
  Baseline: <0.05 | 61 | 72
  Baseline: >=0.05 <0.20 | 9 | 5
  Baseline: >=0.20 <0.40 | 0 | 1
  Baseline: >=0.40 | 0 | 0
  Baseline: Not assessed | 8 | 5
  Day 29: <0.05 | 27 | 27
  Day 29: >=0.05 <0.20 | 1 | 1
  Day 29: >=0.20 <0.40 | 0 | 0
  Day 29: >=0.40 | 0 | 0
  Day 29: Not assessed | 50 | 55
  EoT initial Treatment phase: <0.05 | 62 | 69
  EoT initial Treatment phase: >=0.05 <0.20 | 2 | 2
  EoT initial Treatment phase: >=0.20 <0.40 | 0 | 0
  EoT initial Treatment phase: >=0.40 | 0 | 0
  EoT initial Treatment phase: Not assessed | 14 | 12
  EoT Extension phase: <0.05 | 10 | 11
  EoT Extension phase: >=0.05 <0.20 | 1 | 1
  EoT Extension phase: >=0.20 <0.40 | 0 | 0
  EoT Extension phase: >=0.40 | 0 | 0
  EoT Extension phase: Not assessed | 67 | 71

ADVERSE EVENTS:
Time Frame: Monitoring of AEs, including SAEs, was conducted throughout the study. The Investigator or designee recorded all AEs after informed consent and until the patient's last follow-up visit. The minimum monitoring period was 7 days after first treatment and the maximum period was up to day 92 after first treatment.
Description: Analyses were focused on TEAEs and were performed by primary MedDRA SOC and PT. Patients were counted only once if they had more than one TEAE within a SOC or experienced a PT more than once; when an AE occurs more than once for a patient, the maximum severity and causality was used.
  Data shown refer to Treatment Emergent Adverse Events (TEAEs) only.
Arm/Group | Intralipid® 20% | Smoflipid 20%
All-Cause Mortality (participants affected / at risk) | 1/78 | 1/83
Serious Adverse Events (participants affected / at risk) | 5/78 | 8/83
Other Adverse Events (participants affected / at risk) | 55/78 | 59/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralipid® 20% (N=78) | Smoflipid 20% (N=83)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Candida test positive (Investigations) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralipid® 20% (N=78) | Smoflipid 20% (N=83)
Anemia (Blood and lymphatic system disorders) | 8 (11) | 4 (5)
Anemia neonatal (Blood and lymphatic system disorders) | 17 (20) | 15 (16)
Tachycardia (Cardiac disorders) | 4 (6) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 16 (25) | 15 (27)
Cholestasis (Hepatobiliary disorders) | 9 (9) | 7 (7)
Bilirubin conjugated increased (Investigations) | 7 (8) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 1 (1)
C-reactive protein increased (Investigations) | 7 (7) | 6 (8)
Cardiac murmur (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 11 (12) | 10 (10)
Hematocrit decreased (Investigations) | 5 (6) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 5 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (7)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02579265/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02579265/SAP_001.pdf